CLINICAL TRIAL: NCT02655068
Title: Efficacy of Monitoring Strategies Following Definitive Therapy for Locally Advanced Head and Neck Cancer: A Randomized, Phase III Trial of PET/CT vs. CT Surveillance
Brief Title: Phase III Trial of PET/CT vs. CTSurveilance for Head and Neck Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: due to non-feasibility
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jonas Johnson, Professor and Chair of the Department of Otolaryngology, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UPCI 12-057
Record Dates: First submitted 2015-12-01; First posted 2016-01-13 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck
Keywords: Head and Neck Cancer; Definitive Therapy; Positron Emission Tomography - Computed Tomography (PET/CT); Computed Tomography (CT)
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Computed Tomography (CT) (Other): Patients who undergo primary surgery will have their first study imaging surveillance at 3 months (+/- 30 days) post-surgery. CT surveillance will continue at 6,9,12,18,24 months.
  During years 3-5, or long term follow up, surveillance with history and physical examination will occur every 6 months (+/- 30 days).
  The last protocol-specified imaging will occur at 24 months; during long term follow-up imaging will be conducted per the judgment of the treating physicians, as indicated by the history and physical examination findings.
  Interventions: Other: Computed Tomography (CT)
- PET/CT (Other): Patients who undergo primary radiotherapy will have their first study imaging surveillance at 6 months (+/- 30 days) post radiotherapy. The Positron Emission Tomography - Computed Tomography (PET/CT)surveillance will continue at 9,12,18,24 months.
  During years 3-5, or long term follow up, surveillance with history and physical examination will occur every 6 months (+/- 30 days).
  The last protocol-specified imaging will occur at 24 months; during long term follow-up imaging will be conducted per the judgment of the treating physicians, as indicated by the history and physical examination findings.
  Interventions: Other: PET/CT

INTERVENTIONS:
Other: PET/CT — Patients who undergo primary radiotherapy will have their first study imaging surveillance at 6 months (+/- 30 days) post radiotherapy. The Positron Emission Tomography - Computed Tomography (PET/CT)surveillance will continue at 9,12,18,24 months.
  During years 3-5, or long term follow up, surveillance with history and physical examination will occur every 6 months (+/- 30 days).
  The last protocol-specified imaging will occur at 24 months; during long term follow-up imaging will be conducted per the judgment of the treating physicians, as indicated by the history and physical examination findings.
  Arms: PET/CT
Other: Computed Tomography (CT) — Patients who undergo primary surgery will have their first study imaging surveillance at 3 months (+/- 30 days) post-surgery. CT surveillance will continue at 6,9,12,18,24 months.
  During years 3-5, or long term follow up, surveillance with history and physical examination will occur every 6 months (+/- 30 days).
  The last protocol-specified imaging will occur at 24 months; during long term follow-up imaging will be conducted per the judgment of the treating physicians, as indicated by the history and physical examination findings
  Other Names: CT
  Arms: Computed Tomography (CT)

SUMMARY:
The null hypothesis is that patients screened by PET/CT will not have detection of disease recurrence any earlier than those screened by CT alone. The alternative hypothesis is that PET/CT surveillance will lead to detection of disease recurrence 3 months earlier than CT surveillance. Furthermore, to reject the null hypothesis, earlier detection must be associated with a cause-specific survival improvement of 10%. Primary endpoints will include time from the completion of definitive therapy to diagnosis of recurrent disease, and absolute survival within 3 years after completion of initial therapy. Duration of survival between diagnosis of recurrence and subsequent death will not be a primary endpoint because the investigators expect that PET/CT will offer an opportunity for earlier recognition of recurrence and be subject to lead-time bias. Duration of survival will be measured from completion of primary treatment until death. Note: the presence of residual disease at surgical consolidation does not constitute a recurrence event.

DETAILED DESCRIPTION:
Head and neck cancer (HNC) is the sixth leading incident cancer worldwide with 600,000 cases expected in 2012.1 The vast majority of cases are head and neck squamous cell carcinoma (HNSCC), comprising > 90% of histologies. Despite advances in multimodality therapy for HNSCC, 5-year overall survival (OS) is 40-60%, and has increased only incrementally in the past two decades.2 Improved prognosis is largely attributable to the emerging epidemic of oral human papillomavirus infection (HPV). An increasing proportion of oropharyngeal HNC is driven by oncogenic HPV, rather than the classic risk factors of tobacco and alcohol; HPV etiology is associated with improved survival after conventional treatments.3,4 Most patients with HNC present with locally advanced disease (stage III-IVb), and have associated anatomic deformity due to the primary tumor or neck adenopathy. Intensive multi-modality therapy including surgery, chemotherapy, and radiotherapy is routinely required. The current standard of care for primary nonsurgical management of previously untreated locally advanced (PULA) HNSCC is concurrent cisplatin-radiotherapy (RT), as administered in the sentinel Intergroup trial 0126 5,6. Likewise, the standard of care in the adjuvant management of high risk disease is cisplatin-RT as proven in the Radiation Therapy Oncology Group (RTOG) 95-01 and European Organization for Research and Treatment of Cancer (EORTC) 22931 trials.7,8 Despite curative-intent surgical or non-surgical therapy, approximately half of people will relapse. Unlike most other epithelial malignancies, the dominant pattern of relapse and the driver of HNC-related mortality is locoregional recurrence.9 The vast majority of recurrences occur within the first two years following definitive therapy.

Patient evaluation following completion of definitive therapy for HNC is confounded by anatomic deformity which began with the primary tumor and nodal metastatic disease, and is further compounded by treatment-related effects such as scarring, flap reconstruction, and edema. There currently does not exist an ideal method for surveillance. National Comprehensive Cancer Center Network (NCCN) guidelines call for physical examination and intermittent imaging as required. Clinical trial designs incorporating definitive chemoradiotherapy typically employ a diagnostic, contrast-enhanced CT of the neck every 3 months for 1 year, followed by every 6 months for 1 year, followed by annual evaluations (eg. ECOG 1308; UPCI 07-021). Single-arm prospective studies have suggested that positron emission tomography (PET) with fluorodeoxyglucose (FDG) is more sensitive than CT or physical examination alone for residual or recurrent disease, particularly when conducted with integrated diagnostic CT scan. In these studies, negative PET/CT scans correlated with lower likelihood of residual nodal pathology and improved DFS.12,13 The current practice at the University of Pittsburgh is to employ PET/CT surveillance, in particular following definitive chemoradiotherapy. However, prior investigations have not demonstrated improved salvage or survival outcomes with use of PET/CT surveillance, which is clearly more costly than CT surveillance and may carry morbidity related to increased diagnostic procedures for false-positive findings.

The investigators propose a prospective, randomized phase III trial in patients undergoing definitive therapy for locally advanced Stage III-IVb carcinoma involving the head and neck. This includes primary tumors of the oral cavity, pharynx, and larynx, as well as cancer of the salivary glands and squamous cell carcinoma of the skin. Patients who have realized a clinical complete response to definitive therapy will be randomized to PET/CT vs. CT surveillance, to test the hypothesis that PET/CT surveillance is superior to CT surveillance due to earlier diagnosis of recurrence, more timely and effective salvage, and consequent reduction in HNC mortality. The study intervention will solely be the imaging modality assigned for surveillance. All study patients will otherwise be monitored strictly according to NCCN guidelines, including history and physical examination (and endoscopy where appropriate). Assigned imaging will be conducted at identical intervals. Areas suspicious for recurrence on the basis of history and physical examination, endoscopy or imaging will be biopsied. Therapeutic interventions will be determined by the treatment team, which will include at least one member from medical oncology, radiation oncology, and otolaryngology/head and neck surgery. Patients with recurrent locoregional disease will be offered salvage treatment as indicated by the clinical situation.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed carcinoma arising in the head and neck. Histologies may include squamous cell carcinoma, poorly differentiated carcinoma, carcinoma NOS, basaloid carcinoma, or salivary gland carcinoma (including mucoepidermoid carcinoma, salivary duct carcinoma, adenocarcinoma, and adenoid cystic carcinoma).

  2. Primary site of origin must be one of the following: a) the oral cavity, pharynx, or larynx; b) major or minor salivary gland; c) skin; d) unknown primary site is acceptable in patients with squamous cell carcinoma metastatic to cervical lymph nodes.

  3. Stage III-IVb based upon AJCC 7th edition staging criteria. 4. Serum creatinine ≤ 1.5 mg/dL (most recent within the last three months) 5. The treating multidisciplinary team agrees that the patient has no evidence of disease (NED) after definitive therapy.
  1. Patients who have undergone primary surgery with R0 or R1 resection are eligible to enter the protocol for 6 weeks after the date of definitive surgery. Note: Patients treated with primary surgery will undergo first study surveillance 3 months (+/- 30 days) after the date of definitive surgery.
  2. Patients who have undergone primary radiotherapy (including chemoradiotherapy) must have completed first response assessment 6-14 weeks after completion of radiotherapy. To be eligible, patients must be determined by the multidisciplinary team to without clear evidence of residual disease, without need of surgical consolidation, and appropriate to enter surveillance. Such patients are eligible to enter the surveillance protocol for 6 weeks after the date of first response assessment. Patients requiring surgical consolidation of the primary site and/or neck are eligible following the consolidative surgery, provided benign findings or negative margins were attained. Such patients are eligible to enter the surveillance protocol for 6 weeks after the date of consolidative surgery.

     Note: Patients treated with primary radiotherapy will undergo first study surveillance 6 months (+/-30 days) after completing radiotherapy.

     6. In the case of oropharyngeal primary squamous cell carcinomas, HPV status must be classified per standard of care. HPV(+) disease will be those cases which demonstrate diffuse nuclear and cytoplasmic staining in ≥ 70% tumor cells by p16 immunohistochemistry (IHC).

     7. Age ≥ 18 years 8. Able to provide written, informed consent 9. ECOG Performance Status 0-2

     Exclusion Criteria:
* Severe allergy to iodinated contrast, despite appropriate premedications 2. Presence of gross residual disease after surgical resection 3. Serum creatinine > 1.5 mg/dL 4. Who Type II or III non-keratinizing squamous cell carcinoma of the nasopharynx

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-05; Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Which type of surveillance following definitive therapy for HNC is superior, PET/CT or CT surveillance | 3 years
  All patients will be followed for disease recurrence for at least 3 years after completing primary treatment. The date of documented disease recurrence will be noted and the elapsed time from completion of definitive therapy (surgery or last day of radiotherapy) to recurrence will serve as the co-primary endpoint. A comparison of time to recurrence between the two arms will be conducted only with patients having a documented recurrence. The outcome will be measured using tumor measurements at each follow up scan and documents using RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Johnson, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Center, Pittsburgh, Pennsylvania, United States